CLINICAL TRIAL: NCT06649357
Title: Comparison Between Bipolar Transurethral Resection of the Prostate and Moses Assisted Holmium Laser Enucleation of the Prostate. A Prospective Randomized Multicentric Study
Brief Title: Comparison Between Bipolar Transurethral Resection of the Prostate and Moses Assisted Holmium Laser Enucleation of the Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Ivan Schwartzmann, MD, Principal Investigator, Fundacio Puigvert
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2024 35
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Hyperplasia; Surgery; Endoscopic Anatomical Enucleation of the Prostate (EEAP)
Keywords: Prostate hyperplasia; Surgery; Endoscopic anatomical enucleation of the prostate (EEAP)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Patients who are candidates according to standard medical practice for BPH surgery with a prostate volume ≤ 80 cc measured by urological ultrasound or magnetic resonance imaging (MRI). Surgery will be randomly assigned using MoLEP or Bi-TURP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MoLEP (Active Comparator): Endoscopic Prostate Enucleation Using Moses 2.0 Technology Pulse modulation technology in Moses 2.0applied to Holmium Laser Endoscopic Prostate (MoLEP).
  Interventions: Procedure: MoLEP
- BiTURP (Active Comparator): Bipolar Transurethral Resection of the Prostate
  Interventions: Procedure: BiTURP

INTERVENTIONS:
Procedure: MoLEP — Patients with an indication for surgery for BPH via EEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or BiTURP. A qualified surgeon, having completed their learning curve for endoscopic enucleation (more than 50cases) and possessing experience with both laser types, will perform the surgical procedure.
  Arms: MoLEP
Procedure: BiTURP — Patients with an indication for surgery for BPH viaEEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or BiTURP. A qualified surgeon, having completed their learning curve for endoscopic enucleation (more than 50cases) and possessing experience with both laser types, will perform the surgical procedure.
  Arms: BiTURP

SUMMARY:
Introduction: Multiple studies have demonstrated the superiority of HoLEP in aspects such as transfusión rates or postoperative stay. On the other hand, no differences have been observed in terms of functional outcomes between both techniques, and surgical times reported in different studies tend to be longer for HoLEP. These results likely contribute to TURP, especially with bipolar energy (Bi-TURP), continuing to be considered by many the gold standard for surgical treatment of BPH.

Sofware and hardware upgrades to the Lumenis Pulse 120H. system in 2017, delivered MOSES 2.0, a single-use laser fibre used to perform MOSES augmented HoLEP (MoLEP). MoLEP has shown to be superior in intraoperative outcomes when compared to traditional HoLEP. The availability of new morcellators might also decrease surgical time for HoLEP. This changing landscape for BPH endoscopic surgery deserves a re-evaluation of the differences between Bi-TURP and MoLEP.

Primary Objective: To compare the hospital stay of patients of patients undergoing MoLEP with those undergoing Bi-TURP.

Secondary objectives:

* To compare the surgical time of MoLEP with that of Bi-TURP.
* To compare the bladder catheterization time aCer MoLEP with that of Bi-TURP.
* To compare the postoperative complication rate patients undergoing MoLEP with those undergoing Bi-TURP.
* To compare functional results of patients undergoing MoLEP with those undergoing Bi-TURP.

This study is a prospective multicentric randomized and controlled trial. The study compares two types of BPH surgery without changing standard medical practice.

The study will include patients who are candidates according to standard medical practice for BPH surgery. Patients will be randomized to one of two groups of treatment.

* The MoLEP group will receive surgical treatment with MoLEP.
* The Bi-TURP group will receive surgical treatment with Bi-TURP. Surgical technique and postoperative care will follow standard clinical practice at each participating centre.

DETAILED DESCRIPTION:
Introduction: The evolution of surgery for benign prostatic hyperplasia (BPH) has come a long way since Freyer described his technique of open adenomectomy over 100 years ago. The advancement of instruments and surgical techniques has made surgery increasingly les invasive. Transurethral resection of the prostate (TURP) allowed endoscopic treatment of BPH and it is still regarded by many as the gold-standard for BPH surgical treatment. The application of Holmium laser for endoscopic enucleation of the prostate (HoLEP) in the last 20 years has allowed for the surgical treatment of BPH through an endoscopic approach, practically without limitations in prostate size.

Multiple studies have demonstrated the superiority of HoLEP in aspects such as transfusión rates or postoperative stay. On the other hand, no differences have been observed in terms of functional outcomes between both techniques, and surgical times reported in different studies tend to be longer for HoLEP. These results likely contribute to TURP, especially with bipolar energy (Bi-TURP) continuing to be considered by many the gold standard for surgical treatment of BPH.

However, the available studies often have short follow-up periods, most do not report on the surgeon's experience with HoLEP, and were based on early laser and morcellation technology. Sofware and hardware upgrades to the Lumenis Pulse 120H system in 2017, delivered MOSES 2.0, a single-use laser fibre used to perform MOSES augmented HoLEP (MoLEP). MoLEP has shown to be superior in intraoperative outcomes when compared to traditional HoLEP, resulting in shorter enucleation, haemostasis, and total surgical times for similar energy delivered. The availability of new morcellators might also decrease surgical time for HoLEP. This changing landscape for BPH endoscopic surgery deserves a re-evaluation of the differences between Bi-TURP and MoLEP.

Hypothesis: MoLEP surgery is superior to Bi-TURP in terms of postoperative stay, bladder catheter duration, blood loss and transfusion rate, without significant functional outcomes, and retreatment rate, with no significant differences in surgical time.

Objectives:

Primary Objective: To compare the hospital stay of patients of patients undergoing MoLEP with those undergoing Bi-TURP.

Secondary objectives:

* To compare the surgical time of MoLEP with that of Bi-TURP.
* To compare the bladder catheterization time aCer MoLEP with that of Bi-TURP.
* To compare the postoperative complication rate patients undergoing MoLEP with those undergoing Bi-TURP.
* To compare functional results of patients undergoing MoLEP with those undergoing Bi-TURP.

Study Design: This study is a prospective multicentric randomized and controlled trial. The study compares two types of BPH surgery without changing standard medical practice. The CONSORT guidelines for randomized clinical trials will be followed.

Participants: Patients who are candidates according to standard medical practice for BPH surgery with a prostate volume ≤ 80 cc measured by urological ultrasound or magnetic resonance imaging (MRI).

Intervention: The study will include patients who are candidates according to standard medical practice for BPH surgery. Patients will be randomized to one of two groups of treatment.

* The MoLEP group will receive surgical treatment with MoLEP.
* The Bi-TURP group will receive surgical treatment with Bi-TURP. Surgical technique and postoperative care will follow standard clinical practice at each participating centre.

Surgery and Follow-up Schedule:

* Surgeries will be conducted between November 2024 and April 2025
* Initial 6-month follow-up. Database construction and refinement: 2 months. Statistical analysis: 2 months. Preparation of the final report: 2 months. Completion of the first phase of the study: April 2026.
* Second phase follow-up: 24 months. Database construction and refinement: 2 months. Statistical analysis: 2 months. Preparation of the final report: 2 months. Dissemination of results: 2 months. Completion of the second phase of the study: October 2027
* Third phase follow-up: 5 years. Database construction and refinement: 2 months. Statistical analysis: 2 months. Preparation of the final report: 2 months. Dissemination of results: 2 months. Completion of the third phase of the study: October 2030.

Sample size calculation was calculated based on length of hospital stay. Previous studies indicate that the mean days of hospital stay is around 2,5 days in patients with RTU. The length of hospital stay for patients with MoLEP may be at least 1 day less. Around 10% of patients are treated with antiplatelet agents. In order to perform an analysis according to patients with and without this treatment, the sample size will be increased by 10%. Accepting an alpha risk of 5% and a beta risk of 20% in a two-tailed test, a total of 130 patients are needed (65 in each study group). A common standard deviation of 1 day is assumed. A loss to follow-up rate of 12% has been also estimated.

Statistical Analysis: Qualitative variables will be described with absolute frequencies and percentages. The description of quantitative variables will be performed using the mean, standard deviation (SD), median and quartiles. The Kolmogorov-Smirnov test will be used to assess the normality of distributions.

An initial bivariate intention to treat analysis will be performed in order to analyze potential differences according study groups. The relationship between two qualitative variables will be calculated using the chi-squared test or Fisher's exact test (frequency <5). Quantitative variables will be compared using the Student's t-test (Mann Whitney. For non-normal distributions), analysis of variance [ANOVA] (> 2 categories), linear regression test and Schea's multiple comparisons test. The linear relationship between the quantitative variables will be calculated using Pearson's correlation coefficient or Spearman's rank correlation test (when variable not normally distributed). Changes at the end of follow up in the main outcomes will be analyzed by Wilcoxon nonparametric test in the case of quantitative variables. The McNemar test will be used for the comparison of categorical variables. A backward stepwise linear regression analysis will be performed in order to determine which factors are independently associated to higher length of hospital stay. Study groups and variables with a p value <0.2 in the univariate analysis will be included as independent variables. The results will be described with beta coefficient , 95% confidence interval (CI) and p-values. For all the tests, p-values < 0.05 were considered statistically significant. The statistical package R Studio (V2.5.1) was used for the analyses.

Publications will be made with the results of the study, whether they are positive or negative. There will be at least 3 publication scheduled. This will be the results at 6 months, 2 years, and 5 years of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maximum flow rate < 15 ml/sec before obstructive surgery or with maximum flow rate > 15 ml/sec and urodynamic study showing high-flow obstruction defined as bladder outlet obstruction index > 40.
* Patients with moderate to severe lower urinary tract symptoms (LUTS) according to the International Prostate Symptom Score (IPSS). Score between 8 and 35.
* Patients with a prostate volume between 40 and 80 cc, measured by urological ultrasound or MRI.

Exclusion Criteria:

* History of prior prostatic obstructive or urethral surgery.
* Diagnosis of prostate neoplasia.
* Diagnosis of urothelial neoplasia.
* Lack of flowmetry or IPSS data before surgery.
* Diagnosis or suspicion of hypo/acontractile detrusor before prostatic obstructive surgery.
* Diagnosis or suspicion of neurogenic bladder or neurological disease.
* History of pelvic radiation therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males with an indication for BPH surgery with a prostatic volume >80cc measured by urological ultrasound or magnetic resonance imaging (MRI).
Enrollment: 130 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | From date and time of end of surgery to date and time of hospital discharge assessed up to 1 month
  Variation in length of hospital stay after each procedure. Difference in postoperative hospital stay time between MoLEP and BiTURP. Number of hours in the hospital after the procedure if finished, organized in the following categories: Outpatient procedure (less than 16 hours), 1 day of hospitalization (≤ 24 hours), 2 days of hospitalization (≤ 48 hours), 3 days of hospitalization (≤ 72 hours). Individual length of stay will be recorded).

SECONDARY OUTCOMES:
SURGICAL TIME | Total time of Surgery procedure
  Difference in surgical time between MoLEP and BiTURP in prostates larger than 80 cc.
The bladder catheterization time | Total time of bladder catheterization procedure
  Difference in the bladder catheterization time after MoLEP with that of Bi-TURP
Perioperative complications | From date of surgery to date of the end of follow-up 5 years
  Difference in the incidence of perioperative complications between MoLEP and ThuFLEP. All possible complications will berecorded and classifi ed according to the Clavien- Dindo scale from date of surgery to end of study.
TREATMENT | From date of surgery to date of the end of follow-up 5 years
  Variation in treatment efficacy between groups. Difference in improvement after MoLEP compared to BiTURP
Urinary symptoms | From date of enrollment to date of the end of follow-up 5 years
  Incidence of additional treatment requirement for lower urinary tract symptoms after the treatment. Difference in improvement of urinary symptoms after MoLEP compared to BiTRUP. IPSS questionnaire will be performed in all study visits: Changes in total score and quality of life score before and after surgery will be compared between patients undergoing MoLEP and BiTURP.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Schwartzmann Jochamowitz, MD, Principal Investigator — Fundacio Puigvert
Locations (6):
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Fundacio Puigvert, Barcelona, BARCELONA
  - Hospital Univesitari de Bellvitge, L'Hospitalet de Llobregat, BARCELONA
  - Hospital Universitario Marqués de Valdecillas, Santander, Cantabria
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Río Hortega, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Publications will be made with the results of the study, whether they are positive or negative. There will be at least 3 publications scheduled. This will be the results at 6 months, 2 years, and 5 years of follow up.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available when the study results are published.
Access Criteria: Open

REFERENCES:
- [Background] Stout TE, Borofsky M, Soubra A. A Visual Scale for Improving Communication When Describing Gross Hematuria. Urology. 2021 Feb;148:32-36. doi: 10.1016/j.urology.2020.10.054. Epub 2020 Dec 5. PMID 33285214
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Dowd K, ElMansy H, Sharour W, Kotb A, Shaver C, El Tayeb MM. Wolf Piranha vs Storz Prostate Morcellation Devices: A Retrospective Multi-Institutional Study. J Endourol. 2021 Nov;35(11):1671-1674. doi: 10.1089/end.2020.0541. PMID 34128395
- [Background] Gauhar V, Gilling P, Pirola GM, Chan VW, Lim EJ, Maggi M, Teoh JY, Krambeck A, Castellani D. Does MOSES Technology Enhance the Efficiency and Outcomes of Standard Holmium Laser Enucleation of the Prostate? Results of a Systematic Review and Meta-analysis of Comparative Studies. Eur Urol Focus. 2022 Sep;8(5):1362-1369. doi: 10.1016/j.euf.2022.01.013. Epub 2022 Jan 31. PMID 35105516
- [Background] Zhang Y, Yuan P, Ma D, Gao X, Wei C, Liu Z, Li R, Wang S, Liu J, Liu X. Efficacy and safety of enucleation vs. resection of prostate for treatment of benign prostatic hyperplasia: a meta-analysis of randomized controlled trials. Prostate Cancer Prostatic Dis. 2019 Dec;22(4):493-508. doi: 10.1038/s41391-019-0135-4. Epub 2019 Feb 28. PMID 30816336
- [Background] Kuntz RM, Lehrich K, Ahyai SA. Holmium laser enucleation of the prostate versus open prostatectomy for prostates greater than 100 grams: 5-year follow-up results of a randomised clinical trial. Eur Urol. 2008 Jan;53(1):160-6. doi: 10.1016/j.eururo.2007.08.036. Epub 2007 Aug 28. PMID 17869409
- [Background] Naspro R, Suardi N, Salonia A, Scattoni V, Guazzoni G, Colombo R, Cestari A, Briganti A, Mazzoccoli B, Rigatti P, Montorsi F. Holmium laser enucleation of the prostate versus open prostatectomy for prostates >70 g: 24-month follow-up. Eur Urol. 2006 Sep;50(3):563-8. doi: 10.1016/j.eururo.2006.04.003. Epub 2006 May 2. PMID 16713070
- [Background] Gravas S, Gacci M, Gratzke C, Herrmann TRW, Karavitakis M, Kyriazis I, Malde S, Mamoulakis C, Rieken M, Sakalis VI, Schouten N, Speakman MJ, Tikkinen KAO, Cornu JN. Summary Paper on the 2023 European Association of Urology Guidelines on the Management of Non-neurogenic Male Lower Urinary Tract Symptoms. Eur Urol. 2023 Aug;84(2):207-222. doi: 10.1016/j.eururo.2023.04.008. Epub 2023 May 17. PMID 37202311
- [Background] Freyer PJ. A New Method of Performing Perineal Prostatectomy. Br Med J. 1900 Mar 24;1(2047):698-9. doi: 10.1136/bmj.1.2047.698-a. No abstract available. PMID 20758920